CLINICAL TRIAL: NCT03344666
Title: Adaptive Interventions to Reduce Risky Drinking and Violent Behaviors Among Adolescents
Brief Title: SafERteens M-Coach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Maureen A Walton, Professor, University of Michigan
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: HUM00109156; R01AA024755 (NIH)
Record Dates: First submitted 2017-11-03; First posted 2017-11-17 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Alcohol Drinking; Violence
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- First Treatment (Experimental): Participants will be randomized to first treatment to compare Brief Intervention + Health Coach (Step 1 Treatment BI+HC) to Brief Intervention + Text Messages (Step 1 Treatment BI+TM). Participants in the BI+HC will receive a BI in the ED, followed by weekly sessions with the Health Coach for 4 weeks. Participants in the BI+TM will receive a BI in the ED, followed by daily TMs for 4 weeks.
  Interventions: Behavioral: Step 1 Treatment BI+HC; Behavioral: Step 1 Treatment BI+TM
- Second Treatment for Responders and Non-Responders (Experimental): Beginning in week 5, all participants will be classified as Responders or Non-Responders (based on weekly assessments) and re-randomized.
  Step 2 Treatment Responders: Responders will be randomized to either stay the course or be stepped down. Specifically, participants in the BI+HC will either continue to receive the HC or stepped down to receive a control brochure; participants in the BI+TM will either continue to receive the TM or stepped down to receive a control brochure.
  Step 2 Treatment Non-Responders: Non-Responders will be randomized to either stay the course or be stepped up. Specifically, participants in the BI+HC will either continue to receive the HC or stepped up to receive a HC+; participants in the BI+TM will either continue to receive the TM or stepped up to receive HC.
  Interventions: Behavioral: Step 2 Treatment Responders; Behavioral: Step 2 Treatment Non-Responders

INTERVENTIONS:
Behavioral: Step 1 Treatment BI+HC — Participants in the Brief intervention + Health Coach (BI+HC) will receive a BI in the ED, followed by weekly sessions with the Health Coach for 4 weeks, which will occur by phone or in person. During sessions, the HC will review the prior week's progress, and discuss goals and plans for the following week.
  Arms: First Treatment
Behavioral: Step 1 Treatment BI+TM — Participants in the Brief intervention + Text messages (BI+TM) will receive a BI in the ED, followed by daily TMs for 4 weeks. TM's are tailored based on weekly surveys and focus on motives for alcohol and violence and strategies to reduce involvement.
  Arms: First Treatment
Behavioral: Step 2 Treatment Responders — Participants in the BI+HC assigned to stay the course (e.g., continue to receive the HC) will have 4 more weekly sessions with the HC.
  Participants in the BI+TM assigned to stay the course (e.g., continue to receive the TM) will receive 4 more weeks of TM.
  Participants in the BI+HC or BI+TM assigned to stepped down control will receive a brochure containing community resources.
  Arms: Second Treatment for Responders and Non-Responders
Behavioral: Step 2 Treatment Non-Responders — Participants in the BI+HC assigned to be stepped up will receive HC+, which will consist of weekly sessions as well as on daily TMs from the HC.
  Participants in the BI+HC assigned to stay the course (e.g., continue to receive the HC) will have 4 more weekly sessions with the HC.
  Participants in the BI+TM assigned to be stepped up will receive the HC, which consists of 4 weekly sessions with the HC.
  Participants in the BI+TM assigned to stay the course (e.g., continue to receive the TM) will receive 4 more weeks of TM.
  Arms: Second Treatment for Responders and Non-Responders

SUMMARY:
This study will use a SMART (Sequential, Multiple Assignment Randomized Trial) design to optimize adaptive interventions (AIs) for adolescents reporting alcohol misuse and violent behaviors. The study will test the efficacy of state-of-the-art adaptive intervention delivery approaches (text messaging, remote therapy) for reducing alcohol use and violent behaviors among urban teens. Given the morbidly/mortality associated with alcohol use and violence, this study will have significant impact by using a SMART design to identify the optimal intervention strategy to produce and sustain outcomes among at-risk youth.

DETAILED DESCRIPTION:
The specific aims are to: 1) Compare the efficacy of adaptive interventions (AIs) that begin with BI+TM (brief intervention + text messaging) vs. BI+HC (brief intervention + remote health coach) on reducing alcohol misuse and violent behaviors among youth while in the Emergency Department (ED); and, 2) Identify the most efficacious second-stage strategy post-ED visit for those who initially respond and for those who do not. Specifically, 700 youth (ages 14-20) in the ED screening positive for alcohol use and violent behaviors will be randomly assigned to: BI+TM or BI+HC. After receiving the SafERteens BI in the ED, youth will complete weekly assessments over an 8 week period to tailor intervention content and measure mechanisms of change, with one month determination of participant response (e.g., binge drinking, violence). Responders in each arm will be re-randomized to continued condition (e.g., stay the course or maintenance), or reduced condition (e.g., stepped down). Non-responders will be re-randomized to continued condition (e.g., stay the course or maintenance), or intensified condition (e.g., stepped up). Follow-up assessments will take place at 4 and 8 months post-baseline.

ELIGIBILITY:
Inclusion Criteria:

* patients age 14-20 years presenting to the ED for any reason(except exclusions as noted below)
* past 4 month binge alcohol use and violent behaviors (i.e., physical aggression)
* have a cell phone with texting capabilities and a cell phone plan for texting

Exclusion Criteria:

* patients who do not understand English
* patients deemed unable to provide informed consent due to mental incompetence, incarceration, or medically unstable (abnormal vital signs requiring urgent resuscitation) or
* present for acute suicidal ideation or acute suicide attempt, child abuse, or sexual assault

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Change in Alcohol Consumption | 4 months and 8 months post baseline
  Alcohol consumption will be assessed using the 30-day Timeline Follow-Back (TLFB). The TLFB will capture information on the frequency and quantity of alcohol use including binge drinking, with total consumption calculated.
Change in Physical Violence | 4 months and 8 months post baseline
  Physical violence will be assessed using the 30-day Timeline Follow-Back (TLFB). The TLFB will capture information on the frequency and severity of violent behaviors (e.g. push, shove, slap, kick, punch, weapon/firearm use or carriage etc.), with total violence calculated weighted by severity.

SECONDARY OUTCOMES:
Change in Alcohol Consequences | 4 months and 8 months post baseline
  Alcohol related consequences will be measured using the Young Adult Alcohol Consequences Questionnaire (YAACQ). This study will use a 24-item scale with the following responses (and values):
  0 = None
  1. = 1-2 times
  2. = 3-5 times
  3. = More than 5 times
  The responses will be summed for a total score.
Change in Violence Consequences | 4 months and 8 months post baseline
  Violence related consequences will be assessed using 13 items with following responses (and values):
  0 = None
  1. = 1-2 times
  2. = 3-5 times
  3. = More than 5 times
  These items will assess consequences such as injury, arrest, trouble at school or work, arguments or trouble getting along with friends and/or family members, feeling guilty, unable to stop/desire to fight, and worry or revenge as a result of participant's fighting. Responses are summed to create a total score.

CONTACTS AND LOCATIONS:
Overall Officials: Maureen A Walton, MPH, PhD, Principal Investigator — University of Michigan
Locations (4):
- United States (4):
  - University of Michigan, Ann Arbor, Michigan
  - Ascension St. John Hospital - Emergency Department, Detroit, Michigan
  - Hurley Medical Center - Emergency Department, Flint, Michigan
  - Covenant Healthcare Emergency Care Center, Saginaw, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Walton MA, Carter PM, Seewald L, Ngo Q, Battisti KA, Pearson C, Blow FC, Cunningham RM, Bourque C, Kidwell KM. Adaptive interventions for alcohol misuse and violent behaviors among adolescents and emerging adults in the emergency department: A sequential multiple assignment randomized controlled trial protocol. Contemp Clin Trials. 2023 Jul;130:107218. doi: 10.1016/j.cct.2023.107218. Epub 2023 May 5. PMID 37148999

DOCUMENTS (1):
  • Informed Consent Form (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/66/NCT03344666/ICF_000.pdf